CLINICAL TRIAL: NCT03768154
Title: Prone Positioning and Spontaneous Breathing: a Feasibility Study
Brief Title: Prone Positioning and Spontaneous Breathing
Acronym: PROSE
Status: Unknown | Phase: Phase 1 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Osaka University (Other)
Collaborators: Hospital Rebagliati (Unknown)
Responsible Party: Sponsor
Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: PROSE
Record Dates: First submitted 2018-11-15; First posted 2018-12-07 (Actual); Last update posted 2020-05-15 (Actual); Status verified 2020-05

CONDITIONS: Critical Illness; ARDS
Keywords: spontaneous breathing; prone position; muscle paralysis
MeSH Terms: conditions — Critical Illness | interventions — Supine Position; Prone Position

STUDY DESIGN:
Intervention Model Description: Measurement 1 (Supine + spontaneous effort) , Measurement 2 (Supine + paralysis) , Measurement 3 (Prone + paralysis) , Measurement 4 (Prone + spontaneous breathing)
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- study arm (Experimental): all patients will receive all four intervention in the same sequential method
  Interventions: Procedure: Supine + spontaneous effort; Procedure: Supine + paralysis; Procedure: Prone + paralysis; Procedure: Prone + spontaneous breathing

INTERVENTIONS:
Procedure: Supine + spontaneous effort — without muscle paralysis in supine position
Procedure: Supine + paralysis — administer muscle paralysis in supine position
Procedure: Prone + paralysis — change the patient position from supine to prone with muscle paralysis
Procedure: Prone + spontaneous breathing — cease the paralysis in supine position

SUMMARY:
Spontaneous breathing during mechanical ventilation has been recommended in patients with ARDS and is currently used. in part because oxygenation is better and there is a lower risk of diaphragm dysfunction due to disuse. The other approach to minimizing lung injury from spontaneous effort is the use of neuromuscular blockade; an early and short term (48 hours) of neuromuscular blockade in patients with severe ARDS has been shown to decrease inflammation and to improve survival. The investigators propose a pilot study to test the feasibility and the physiological effects of allowing spontaneous breathing in the prone position in patients with ARDS.

DETAILED DESCRIPTION:
The multi-center feasibility study will enroll 12 adult ARDS patients from the Intensive Care Units (ICUs) in Japan and Peru. Informed consent will be obtained from the patient or legally authorized substitute decision maker. Moderate-to-severe ARDS patients who are planned to turn to prone positioning, based on the attending physician's decisions will be included. Prior to initiating the protocol, patients will be sedated deeply with sedatives and/or opioids. Ventilator settings, physiological data, esophageal pressure and diaphragm activity will be recorded and physiological measurements will be collected for 5 minutes in supine (Measurement 1: Supine + spontaneous effort) . Patients will be paralyzed with a continuous infusion of rocuronium, and Measurement 2 (Supine + paralysis) will be recorded. The critical care team in the ICU change the position from supine to prone. After waiting for at least 1 hour in prone positioning, Measurement 3 (Prone + paralysis) will be recorded. Continuous infusion of rocuronium will be gradually decreased (and can be terminated) until spontaneous breathing will be observed without reaching an excessive level. The presence of spontaneous breathing will be evaluated by the negative swing of esophageal pressure, and Measurement 5 (Prone + spontaneous breathing) will be recorded.

ELIGIBILITY:
Inclusion Criteria:

* Patients ≧ 18 years old
* Patients with moderate-to-severe ARDS as per the Berlin definition
* Patients with esophageal balloon manometry
* Patients planned to turn to prone positioning, based on the attending physician's decisions

Exclusion Criteria:

* Contraindication for prone positioning, referring to a previous randomized clinical trial

  1. Intracranial pressure >30 mm Hg or cerebral perfusion pressure <60 mmHg
  2. Massive hemoptysis requiring an immediate surgical or interventional radiology procedure
  3. Tracheal surgery or sternotomy during the previous 15 days
  4. Serious facial trauma or facial surgery during the previous 15 days
  5. Cardiac pacemaker inserted in the last 2 days
  6. Unstable spine, femur, or pelvic fractures
* Major hemodynamic instability:

Mean arterial pressure lower than 60 mm Hg despite adequate fluid resuscitation and two vasopressors or increase of vasopressor dose by 30% in the previous 6 hours.

* Contraindication to EIT electrode placement Burns, chest wall bandaging limiting electrode placement, pacemaker
* Clinical judgement of the attending physician against proning and/or spontaneous breathing

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 12 (Estimated)
Dates: Start 2019-03-01 (Actual); Primary Completion 2020-05-08 (Actual); Study Completion 2021-03-31 (Estimated)

PRIMARY OUTCOMES:
spontaneous breathing | Through study completion (up to 24 hours)
  The intensity of spontaneous breathing during supine vs. prone estimated by an esophageal manometry

SECONDARY OUTCOMES:
inflammatory cytokines | Through study completion (up to 24 hours)
  IL-6 levels
Trans-pulmonary pressure | Through study completion (up to 24 hours)
  Trans-pulmonary pressure
electrical activity of diaphragm | Through study completion (up to 24 hours)
  electrical activity of diaphragm
gas exchange | Through study completion (up to 24 hours)
  gas exchange

CONTACTS AND LOCATIONS:
Overall Officials: Takeshi Yoshida, PhD, Principal Investigator — Osaka University
Locations (1):
- Osaka University Hospital, Suita, Osaka, Japan

IPD SHARING:
Plan to Share IPD: No